CLINICAL TRIAL: NCT00534352
Title: A Multicenter Study to Evaluate the Pharmacokinetic Profile and Safety of TMC125 Plus Tenofovir DF/Emtricitabine All Dosed Once Daily With and Without Darunavir (PREZISTA™)/ Ritonavir Once Daily in Antiretroviral naïve HIV-1 Infected Subjects
Brief Title: A Study to Evaluate the Pharmacokinetic Profile (How the Body Absorbs, Distributes, Metabolizes and Eliminates a Drug) of TMC125 Plus Tenofovir/Emtricitabine Once Daily With or Without Darunavir/r Once Daily in Antiretroviral (ARV) Naive HIV-1 Patients (Patients Have Never Received ARV Treatment).
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tibotec, Inc (Industry)
Collaborators: Tibotec Therapeutics, a Division of Ortho Biotech Products, L.P., USA (Industry)
Responsible Party: Vice President Clinical Affairs, Tibotec Therapeutics Clinical Affairs, a Division of Ortho Biotech Clinical Affairs, LLC
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR014485; TMC125HIV2032
Record Dates: First submitted 2007-09-21; First posted 2007-09-24 (Estimated); Results first posted 2010-04-12 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-03

CONDITIONS: HIV-1 Infection
Keywords: HIV; AIDS; Immunodeficiency Virus, Human; PREZISTA; darunavir; TMC114; TMC125; Protease Inhibitor; Non-Nucleoside Reverse Transcriptase Inhibitor; Truvada; Treatment Naive
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — etravirine; Darunavir; Ritonavir

ARMS (1):
- 001 (Experimental): TMC125; darunavir; ritonavirTMC125 400mg once daily for 4 weeks; Darunavir-800mg once daily for 48 weeks; Ritonavir-100mg once daily for 48 weeks
  Interventions: Drug: TMC125; darunavir; ritonavir

INTERVENTIONS:
Drug: TMC125; darunavir; ritonavir — TMC125 400mg once daily for 4 weeks; Darunavir-800mg once daily for 48 weeks; Ritonavir-100mg once daily for 48 weeks

SUMMARY:
The purpose of this study is to determine the pharmacokinetic profile of TMC125 400mg with tenofovir DF/emtricitabine FDC (fixed dose combination) 300/200mg all dosed once daily with and without darunavir/ritonavir 800/100 mg once daily in HIV-1 infected, antiretroviral (ARV) naÃ-ve patients (patients who have never received ARV treatment).

DETAILED DESCRIPTION:
This is a multi-center, open-label (doctors and patients know which drug is being given), Phase IIa clinical trial to evaluate the pharmacokinetic (PK) profile, safety and tolerability of TMC125 dosed once daily with tenofovir/emtricitabine with and without darunavir/ritonavir in antiretroviral naive HIV-1 infected patients. There will be an optional open-label extension phase to evaluate effectiveness, safety and tolerability of continued tenofovir/emtricitabine with darunavir/ritonavir all dosed once daily for 48 weeks. This study will be conducted in the United States at up to 5 sites where 20 patients will initially receive TMC125 400mg with tenofovir DF/emtricitabine FDC 300/200 mg all dosed once daily for 14 days. On Day 15, a blood sample will be obtained and intensive TMC125 pharmacokinetic (PK) values and fasting lipids (check of total cholesterol, direct LDL, HDL, triglycerides) following a 10 hour fast (no eating) will be assessed. Patients will then add darunavir / ritonavir 800/100 mg once a day to the regimen for Days 15 - 29. On Day 29 intensive PK sampling for TMC125, darunavir and ritonavir will be performed and fasting lipids will be evaluated. On Day 29, patients will discontinue TMC125 and continue darunavir/ritonavir 800/100 mg and tenofovir DF/emtricitabine FDC 300/200 mg all dosed once daily. On Day 43, fasting lipids will be assessed. At this point, patients may enter the optional open-label extension phase of the study and continue treatment with darunavir/ritonavir 800mg/100 mg and tenofovir DF/emtricitabine FDC 300/200mg all dosed once daily through 48 total weeks of treatment. The study will consist of a total of 8 visits including 2 intensive PK visits. Within 4 weeks after the Screening Visit, the study site should have received all data to determine a patient's eligibility for the study. The Baseline Visit (Day 1) will be followed by a study visit on Day 8. An intensive PK visit will occur on Day 15. After modification of therapy on Day 15, a study visit will occur on Day 22. A second intensive PK visit will occur on Day 29. On Day 43 a study visit will occur at which point study therapy will be discontinued unless the patient elects to continue in the optional open label extension phase of the study. Patients electing to continue in the open-label extension will have 4 additional study visits at Week 12, 24, 36 and 48. All patients will be asked to return for a 4-week follow-up visit after the completion of study treatment.

During the treatment period, the patient will be seen at regular visits during which the investigator will assess the patient's medical condition, any Adverse Events and study drug compliance. Laboratory evaluations for effectiveness and safety will be done at regular visits as well as blood pressure monitoring. All patients will receive TMC125 400 mg orally (by mouth) once daily. Tenofovir DF 300mg/emtricitabine 200mg will be dosed once daily orally as the fixed dose combination. Darunavir/ritonavir will be dosed 800/100 mg orally once daily. All doses should be administered following a meal.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV-1 infection
* Naive to antiretroviral therapy (never received antiretroviral therapy prior to study)
* In the opinion of the investigator, have an indication for antiretroviral therapy
* Able to comply with the protocol requirements

Exclusion Criteria:

* No previous or current use of antiretroviral medications (ARVs) for the treatment of HIV infection or hepatitis B/C infection with anti-HIV activity
* No evidence of antiretroviral resistance on current or past resistance assays
* No chronic hepatitis B and/or C co-infection
* No grade 3 or 4 laboratory abnormality as defined by National Institute of Allergy and Infectious Diseases Division of Acquired Immunodeficiency Syndrome (DAIDS) grading tables, or a calculated creatinine clearance (CLCr) < 50 mL/min.
* No known diabetes mellitus or hyperlipidemia requiring lipid-lowering therapy
* No acute viral hepatitis including, but not limited to A, B, or C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2008-01; Primary Completion 2008-05 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec, Inc. Clinical Trial, Study Director — Tibotec, Inc

REFERENCES:
- [Derived] DeJesus E, Lalezari JP, Osiyemi OO, Ruane PJ, Ryan R, Kakuda TN, Witek J. Pharmacokinetics of once-daily etravirine without and with once-daily darunavir/ritonavir in antiretroviral-naive HIV type-1-infected adults. Antivir Ther. 2010;15(5):711-20. doi: 10.3851/IMP1562. PMID 20710052

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The 42-day open-label main treatment phase of this trial was conducted from 10 December 2007 to 27 May 2008. Four investigators from the US participated in this multicenter trial. A total of 35 subjects were screened and of these, 23 subjects entered the trial and started the first treatment phase
Groups:
- TDF/FTC +/- TMC125 +/- DRV/Rtv: In the first part of the trial (Days 1-14), all subjects received TMC125 400 mg once daily (qd) in combination with fixed dose combinations (FDC) of tenofovir disoproxil (TDF)/emtricitabine (FTC) 300/200 mg qd(Truvada®) for 14 days (Treatment A: TMC125 + TDF/FTC ). On Day 14, 24-hour intensive TMC125 pharmacokinetic sampling took place and fasting lipids were assessed.
  In the second part of the trial (Days 15-28) darunavir (DRV)/ritonavir (rtv) 800/100 mg qd was added to the regimen (Treatment B: TMC 125 + TDF/FTC + DRV/rtv). On Day 28, 24-hour intensive pharmacokinetic sampling for TMC125, DRV and ritonavir took place and fasting lipids were assessed.
  In the third part of the trial (Day 29-42), TMC125 was discontinued and subjects received treatment with DRV/rtv 800/100 mg q.d. and TDF/FTC FDC 300/200 mg qd (Treatment C: DRV/rtv + TDF/FTC).On Day 42, fasting lipids were assessed.
  Subjects discontinued or entered the optional open-label extension period DRV/rtv + TDF/FTC.
Period: Treatment A: TMC125 + TDF/FTC
Arm/Group | TDF/FTC +/- TMC125 +/- DRV/Rtv
Started | 23
Completed | 21
Not Completed | 2
Not completed — Physician Decision | 1
Not completed — Lost to Follow-up | 1
Period: Treatment B: TMC125 + TDF/FTC + DRV/Rtv
Arm/Group | TDF/FTC +/- TMC125 +/- DRV/Rtv
Started | 21
Completed | 21
Not Completed | 0
Period: Treatment C: DRV/Rtv + TDF/FTC
Arm/Group | TDF/FTC +/- TMC125 +/- DRV/Rtv
Started | 21
Completed | 20
Not Completed | 1
Not completed — Physician Decision | 1
Period: Optional Extension: DRV/Rtv + TDF/FTC
Arm/Group | TDF/FTC +/- TMC125 +/- DRV/Rtv
Started | 18
Completed | 14
Not Completed | 4
Not completed — Physician Decision | 1
Not completed — Lost to Follow-up | 2
Not completed — Pregnancy | 1

BASELINE CHARACTERISTICS:
Arm/Group | TDF/FTC +/- TMC125 +/- DRV/Rtv
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.87 (13.264)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 20
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 9
  Caucasian / White | 9
  Hispanic | 5
Region of Enrollment [Number; unit: participants]
  United States | 23
CYP2C19 Genotyping [Number; unit: participants] — There are 21 participants with genotyping data.
  participants
    CYP2C19*1/CYP2C19*1 : Normal Phenotype | 5
    CYP2C19*1/CYP2C19*17 : Rapid Phenotype | 5
    CYP2C19*1/CYP2C19*2 : Intermediate Phenotype | 7
    CYP2C19*17/CYP2C19*17 : Ultrarapid Phenotype | 1
    CYP2C19*17/CYP2C19*2 : Normal Phenotype | 2
    CYP2C19*2/CYP2C19*2 : Poor Phenotype | 1
    No data | 2
CYP2C9 Genotyping [Number; unit: participants] — There are 21 participants with genotyping data.
  participants
    CYP2C9*1/CYP2C1*1 : Normal Phenotype | 19
    CYP2C9*1/CYP2C1*3 : Intermediate Phenotype | 2
    No data | 2
Family History Related to Skin Disease [Number; unit: participants]
  No | 18
  Yes | 5
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 26.33 (4.629)
Height [Mean (Standard Deviation); unit: cm] | 172.73 (8.405)
Weight [Mean (Standard Deviation); unit: kg] | 78.58 (13.711)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Contributing to the Pharmacokinetic (PK) Evaluations: Cmin, Cmax, AUC24 & Css,av
Description: At visit Days 14 & 28, samples were collected pre-dose and at 1, 2, 3, 4, 6, 9, and 12 hours post-dose. An additional sample was taken at 24 hours (Day 15 or 29 as applicable) post-dose.
Time Frame: 6 weeks
Population: Intention To Treat (ITT) population
Measure: Number; unit: participants
Groups:
- Treatment A: TMC125 + TDF/FTC: Treatment A: TMC125 + TDF/FTC.
- Treatment B: TMC125 + TDF/FTC + DRV/Rtv: Treatment B: TMC125 + TDF/FTC + DRV/rtv.
Arm/Group | Treatment A: TMC125 + TDF/FTC | Treatment B: TMC125 + TDF/FTC + DRV/Rtv
Number analyzed (Participants) | 23 | 21
participants | 23 | 21
Statistical Analysis 1: Comparison: Treatment A: TMC125 + TDF/FTC vs Treatment B: TMC125 + TDF/FTC + DRV/Rtv; Previous studies showed that the intrasubject variability on the log transformed Cmax and AUC12h of TMC125 was less than or equal to 40%. Based on this and with complete data on 20 patients, the 90% CI of the true ratio of the means was expected to be contained within 81-124% of the observed ratio of the means; Test type: Non-Inferiority or Equivalence — Equivalence was shown for Cmin as the 90% confidence intervals (CI) of the LSmean ratio was within the 80-125% limits; Mixed Models Analysis (Cmin) — No p-values; The linear mixed effects model was controlled for treatment as fixed effects, and subject as a random effect; Least Square (LS) mean ratio = 95.47, 90% CI [82.77 to 110.1] — The results are for the mean ratio of Cmin. Numerator: Treatment B Denominator: Treatment A
Statistical Analysis 2: Comparison: Treatment A: TMC125 + TDF/FTC vs Treatment B: TMC125 + TDF/FTC + DRV/Rtv; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Equivalence was shown for Cmax as the 90% confidence intervals (CI) of the LSmean ratio was within the 80-125% limits; Mixed Models Analysis (Cmax) — No p-values; The linear mixed effects model was controlled for treatment as fixed effects, and subject as a random effect; Least Square (LS) mean ratio = 102.6, 90% CI [92.91 to 113.3] — The results are for the mean ratio of Cmax. Numerator: Treatment B Denominator: Treatment A
Statistical Analysis 3: Comparison: Treatment A: TMC125 + TDF/FTC vs Treatment B: TMC125 + TDF/FTC + DRV/Rtv; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Equivalence was shown for AUC24 as the 90% confidence intervals (CI) of the LSmean ratio was within the 80-125% limits; Mixed Models Analysis (AUC24) — No p-values; The linear mixed effects model was controlled for treatment as fixed effects, and subject as a random effect; LS means of ratios = 98.97, 90% CI [89.23 to 109.8] — The results are for the mean ratio of AUC24. Numerator: Treatment B Denominator: Treatment A
Statistical Analysis 4: Comparison: Treatment A: TMC125 + TDF/FTC vs Treatment B: TMC125 + TDF/FTC + DRV/Rtv; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Equivalence was shown for Css,av as the 90% confidence intervals (CI) of the LSmean ratio was within the 80-125% limits; Mixed Models Analysis (Css,av) — No p-values; The linear mixed effects model was controlled for treatment as fixed effects, and subject as a random effect; Least Square (LS) mean ratio = 99.30, 90% CI [89.39 to 110.3] — The results are for the mean ratio of Css,av. Numerator: Treatment B Denominator: Treatment A

2. Secondary Outcome: Number of Participants With Treatment-Emergent Graded Laboratory Abnormalities (Worst Grade): Glucose-Hyperglycemia
Description: Number of Participants with Treatment-Emergent Graded Laboratory Abnormalities (Worst Grade): Glucose-Hyperglycemia.
  Worst Grade is based on the National Institute of Allergy and Infectious Diseases Division of Acquired Immunodeficiency Syndrome (DAIDS) toxicity grading scale, 0,1,2,3,4 and 5 : None, Mild, Moderate, Severe, Life-threatening and Death.
Time Frame: Day 1 through 42 and Week 48
Population: ITT
Measure: Number; unit: participants
Groups:
- Treatment A: TMC125 + TDF/FTC
- Treatment B: TMC125 + TDF/FTC + DRV/rtv
- Treatment C; Optional Extension: DRV/rtv + TDF/FTC
Arm/Group | Treatment A | Treatment B | Treatment C | Optional Extension
Number analyzed (Participants) | 21 | 21 | 20 | 18
participants
  Grade 1 | 1 | 2 | 0 | 2
  Grade 2 | 1 | 0 | 1 | 1

3. Secondary Outcome: Number of Participants With Treatment-Emergent Graded Laboratory Abnormalities (Worst Grade): Glucose- Hypoglycemia
Description: Number of participants with Treatment-Emergent Graded Laboratory Abnormalities (Worst Grade): Glucose- Hypoglycemia.
  Worst Grade is based on the DAIDS toxicity grading scale 0-5: No Toxicity-Death.
Time Frame: Day 1 through 42 and Week 48
Population: ITT
Measure: Number; unit: participants
Arm/Group | Treatment A | Treatment B | Treatment C | Optional Extension
Number analyzed (Participants) | 21 | 21 | 20 | 18
participants
  Grade 1 | 0 | 2 | 0 | 1
  Grade 2 | 0 | 1 | 0 | 0

4. Secondary Outcome: Number of Participants With Treatment-Emergent Non-Graded Laboratory Abnormalities(Worst Abnormality): Glucose- Insulin
Description: Number of participants with Treatment-Emergent Non-Graded Laboratory Abnormalities(Worst Abnormality): Glucose- Insulin.
  Normal Range: 3.0 - 27.0 ulU/mL
Time Frame: Day 1 through 42 and Week 48
Measure: Number; unit: participant
Arm/Group | Treatment A | Treatment B | Treatment C | Optional Extension
Number analyzed (Participants) | 21 | 21 | 19 | 16
participant
  Below 3.0 ulU/mL | 1 | 2 | 1 | 1
  Above 27.0 ulU/mL | 1 | 3 | 2 | 3

5. Secondary Outcome: Number of Participants With Treatment-Emergent Graded Laboratory Abnormalities (Worst Grade): Lipids- Total Cholesteral
Description: Number of participants with Treatment-Emergent Graded Laboratory Abnormalities (Worst Grade): Lipids- Total Cholesteral.
  Worst Grade is based on the DAIDS toxicity grading scale, 0-5 : No Toxicity-Death.
Time Frame: Day 1 through 42 and Week 48
Population: ITT
Measure: Number; unit: participants
Arm/Group | Treatment A | Treatment B | Treatment C | Optional Extension
Number analyzed (Participants) | 21 | 20 | 20 | 7
participants
  Grade 1 | 0 | 0 | 2 | 1
  Grade 2 | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Treatment-Emergent Non-Graded Laboratory Abnormalities(Worst Abnormality): Lipids- High-density Lipoprotein (HDL)
Description: Number of participants with Treatment-Emergent Non-Graded Laboratory Abnormalities(Worst Abnormality): Lipids- High-density lipoprotein (HDL).
  Normal Range:
  40 - 59 mG/dL 1.03 - 1.53 mmol/L
Time Frame: Day 1 through 42 and Week 48
Population: ITT
Measure: Number; unit: participants
Arm/Group | Treatment A | Treatment B | Treatment C | Optional Extension
Number analyzed (Participants) | 14 | 15 | 15 | 7
participants
  Below 40 mG/dL (1.03 mmol/L) | 4 | 8 | 6 | 2
  Above 59 mG/dL (1.53 mmol/L) | 0 | 0 | 0 | 1

7. Secondary Outcome: Number of Participants With Treatment-Emergent Graded Laboratory Abnormalities(Worst Grade): Lipids- Low-density Lipoprotein (LDL) Direct
Description: Number of participants with Treatment-Emergent Graded Laboratory Abnormalities(Worst Grade): Lipids- Low-density lipoprotein (LDL) Direct.
  Worst Grade is based on the DAIDS toxicity grading scale, 0-5 : No Toxicity-Death.
Time Frame: Day 1 through 42 and Week 48
Population: ITT
Measure: Number; unit: participants
Arm/Group | Treatment A | Treatment B | Treatment C | Optional Extension
Number analyzed (Participants) | 21 | 20 | 20 | 7
participants
  Grade 1 | 0 | 0 | 1 | 1
  Grade 2 | 0 | 0 | 1 | 1

8. Secondary Outcome: Number of Participants With Treatment-Emergent Graded Laboratory Abnormalities(Worst Grade): Lipids- Triglycerides
Description: Number of participants with Treatment-Emergent Graded Laboratory Abnormalities(Worst Grade): Lipids- Triglycerides.
  Worst Grade is based on the DAIDS toxicity grading scale, 0-5 : No Toxicity-Death.
Time Frame: Day 1 through 48 and Week 48
Population: ITT
Measure: Number; unit: participants
Arm/Group | Treatment A | Treatment B | Treatment C | Optional Extension
Number analyzed (Participants) | 20 | 19 | 20 | 7
participants
  Grade 1 | 0 | 0 | 0 | 0
  Grade 2 | 0 | 0 | 0 | 0

9. Secondary Outcome: Virologic Response < 50 HIV-1 RNA Copies/mL (ITT-Observed Case)
Description: Virologic Response < 50 HIV-1 RNA Copies/mL (ITT-Observed Case).
Time Frame: Day 8, 14, 22, 28, 42 and Week 48
Population: ITT
Measure: Number; unit: participants
Arm/Group | TDF/FTC +/- TMC125 +/- DRV/Rtv
Number analyzed (Participants) | 23
participants
  Day 8 (n=19) | 0
  Day 14 (n=21) | 3
  Day 22 (n=19) | 4
  Day 28 (n=20) | 6
  Day 42 (n=20) | 7
  Week 48 (n=13) | 10

10. Secondary Outcome: Log10 Viral Load (HIV-1 RNA Copies/mL): Mean Changes From Baseline(ITT-Observed Case)
Description: Log10 Viral Load (HIV-1 RNA copies/mL): Mean Changes From Baseline(ITT-Observed Case).
Time Frame: Baseline, Day 8, 14, 22, 28 & 42 and Week 48
Population: ITT (Observed)
Measure: Mean (Standard Error); unit: copies/mL
Arm/Group | TDF/FTC +/- TMC125 +/- DRV/Rtv
Number analyzed (Participants) | 23
copies/mL
  Baseline (n=23) | 4.19 (0.157)
  Day 8 (n=19) | -1.41 (0.094)
  Day 14 (n=21) | -1.71 (0.090)
  Day 22 (n=19) | -1.77 (0.094)
  Day 28 (n=20) | -1.86 (0.123)
  Day 42 (n=20) | -2.04 (0.127)
  Week 48 (n=13) | -2.30 (0.237)

11. Secondary Outcome: CD4+ Cell Count (x 10^6 Cell/L): Baseline and Median Changes From Baseline (ITT-Observed Case)
Description: CD4+ Cell Count (x 10^6 cell/L): Baseline and Median Changes From Baseline (ITT-Observed Case).
Time Frame: Baseline, Day 8, 14, 22, 28 & 42 ans Week 48
Measure: Median (Full Range); unit: x 10^6 cell/L
Arm/Group | TDF/FTC +/- TMC125 +/- DRV/Rtv
Number analyzed (Participants) | 23
x 10^6 cell/L
  Baseline (n=23) | 403.0 [144.0 to 895.0]
  Day 8 (n=20) | 45.5 [-126.0 to 209.0]
  Day 14 (n=20) | 94.0 [-78.0 to 426.0]
  Day 22 (n=20) | 59.0 [-184.0 to 251.0]
  Day 28 (n=21) | 62.0 [-170.0 to 329.0]
  Day 42 (n=19) | 56.0 [-221.0 to 472.0]
  Week 48 (n=14) | 160.0 [-124.0 to 411.0]

12. Secondary Outcome: CD4+ Cell Count (Percent): Baseline and Median Changes From Baseline (ITT-Observed Case)
Time Frame: Baseline, Day 8, 14, 22, 28 & 42 and Week 48
Population: ITT (Observed)
Measure: Median (Full Range); unit: Percent Change from Baseline
Arm/Group | TDF/FTC +/- TMC125 +/- DRV/Rtv
Number analyzed (Participants) | 23
Percent Change from Baseline
  Baseline (n=23) | 26.2 [11.4 to 48.3]
  Day 8 (n=20) | 0.1 [-7.7 to 8.1]
  Day 14 (n=20) | 4.2 [-3.5 to 10.5]
  Day 22 (n=20) | 1.8 [-4.5 to 7.9]
  Day 28 (n=21) | 3.0 [-0.9 to 11.2]
  Day 42 (n=19) | 4.2 [-2.7 to 14.4]
  Week 48 (n=14) | 3.8 [-0.2 to 11.5]

ADVERSE EVENTS:
Time Frame: Baseline, Day 8, 14, 22, 28, 42 and Week 48
Arm/Group | Treatment A | Treatment B | Treatment C | Optional Extension
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/21 | 0/21 | 1/18
Other Adverse Events (participants affected / at risk) | 10/23 | 9/21 | 4/21 | 13/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A (N=23) | Treatment B (N=21) | Treatment C (N=21) | Optional Extension (N=18)
Burkitt's Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A (N=23) | Treatment B (N=21) | Treatment C (N=21) | Optional Extension (N=18)
Acne Cystic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Anogenital Dysplasia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1
Areflexia (Nervous system disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Blood Urine Present (Investigations) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1
Bronchitis Chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Conjunctival Haemorrhage (Eye disorders) | 0 | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Dermatitus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 1 | 3
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 1
Drug Exposure During Pregnancy (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Fatigue (General disorders) | 1 | 2 | 0 | 0
Folliculitis (Infections and infestations) | 1 | 1 | 0 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 1
Intracranial Hypotension (Nervous system disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 4 | 0 | 2
Oral Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Sinus Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Syphilis (Infections and infestations) | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 1 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If TTCA does not publish within 12 months after study conclusion or after TTCA confirms there will be no multicenter publication, Institution may publish their results from their site individually, provided TTCA has 60 day review for confidentiality and additional 60 day delay for patent application.